CLINICAL TRIAL: NCT02677779
Title: A Randomised, Open Label, Controlled Clinical Study to Evaluate the Efficacy and Safety of CO2-Laser Treatment in Patients With Diabetic Infected Foot Ulcers
Brief Title: CO2-Laser Treatment in Patients With Diabetic Infected Foot Ulcers
Acronym: DULCIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Edoardo Mannucci, Director, Diabetology, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPE 15.161
Record Dates: First submitted 2016-02-03; First posted 2016-02-09 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CO2 laser (Experimental): Ulcer debridement with laser-CO2 (DEKA SmartXide2 c80-El.En, Florence Italy)
  Interventions: Procedure: CO2 laser
- Traditional surgery (Active Comparator): Ulcer debridement with traditional surgery
  Interventions: Procedure: traditional surgery

INTERVENTIONS:
Procedure: CO2 laser — Single session of CO2 laser debridement
  Arms: CO2 laser
Procedure: traditional surgery — Single session of traditional debridement
  Arms: Traditional surgery

SUMMARY:
The study is aimed at comparing debridement either with CO2 laser or traditional surgery in patients with infected diabetic foot ulcers. The principal endpoint is bacterial load immediately after treatment.

DETAILED DESCRIPTION:
The present study is designed to assess the antimicrobial effect of a single CO2 laser beam (DEKA SmartXide2 c80-El.En, Florence Italy) in the treatment of diabetic infected foot ulcers. CO2 laser debridement will be compared with standard surgical care. The primary efficacy endpoint will be the reduction of bacterial load between pre- and immediately after debridement. Secondary endpoints will be adverse events and pain during treatment. Two bacterial sample with a flocked nylon swab will be collected before and after debridement.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes
* Infected foot ulcer (with clinical signs of infection)
* Ulcer area between 0.5 and 150 cm2
* More than 50% of ulcer area covered by fibrin and/or necrosis
* Texas score <3

Exclusion Criteria:

* Need for revascularization
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Mannucci, MD, Principal Investigator — University of Florence

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CO2 Laser | Traditional Surgery
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CO2 Laser | Traditional Surgery | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (11.1) | 76.8 (8.6) | 71.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  Italy | 10 | 10 | 20
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 25.6 (7.0) | 30.8 (8.2) | 28.2 (7.5)
Diabetes duration [Mean (Standard Deviation); unit: years] | 13.7 (12.1) | 20.3 (10.5) | 17.1 (11.2)
HbA1c [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 6.6 (1.0) | 7.4 (1.4) | 7.0 (1.3)
Duration of ulcer [Mean (Standard Deviation); unit: months] | 5.6 (5.3) | 3.3 (3.4) | 4.6 (4.3)
Ulcer area [Mean (Standard Deviation); unit: cm^2] | 2.0 (1.7) | 2.7 (2.8) | 2.3 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Load
Description: Percent change in bacterial colonies from baseline.
Time Frame: Percent change in bacterial colonies from baseline. Variation from baseline and immediately after the end of procedure.
Population: Per-protocol analysis: patients with no detectable bacterial load at baseline were excluded.
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | CO2 Laser | Traditional Surgery
Number analyzed (Participants) | 8 | 8
Percent change from baseline | -99.9 [-100 to -90] | -50.0 [-96.0 to 0]

2. Secondary Outcome: Pain: Scores of Brief Pain Inventory
Description: Scores of Brief Pain Inventory. Scale ranges: from 0 to 10. 0 = No pain; 10= Pain as bad as you can imagine.
Time Frame: During procedure.
Population: ITT analysis: patients with no detectable bacterial load at baseline were included.
Measure: Median (Inter-Quartile Range); unit: cm for a VAS scale.
Arm/Group | CO2 Laser | Traditional Surgery
Number analyzed (Participants) | 10 | 10
cm for a VAS scale. | 0 [0 to 1.5] | 1.0 [0 to 3.7]

3. Secondary Outcome: Fibrin: Percent of Ulcer Area Covered by Fibrin
Description: Percent change of ulcer area covered by fibrin from baseline to immediately after the end of procedure
Time Frame: Baseline and immediately after the end of procedure
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | CO2 Laser | Traditional Surgery
Number analyzed (Participants) | 10 | 10
Percent change from baseline | -83.1 [-91.9 to -75.9] | -42.9 [-61.7 to -30.3]

4. Secondary Outcome: Granulation: Percent of Ulcer Area Covered by Granulation.
Description: Percent change of ulcer area covered by granulation from baseline to immediately after the end of procedure.
Time Frame: Baseline and immediately after procedure
Population: ITT analysis: patients with no detectable bacterial load at baseline were included.
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | CO2 Laser | Traditional Surgery
Number analyzed (Participants) | 10 | 10
Percent change from baseline | 307.7 [164.8 to 932.8] | 230.4 [125.4 to 855.4]

5. Secondary Outcome: Bleeding: Proportion of Patients With Bleeding Necessitating Haemostasis
Description: proportion of patients with bleeding necessitating haemostasis
Time Frame: during procedure
Population: ITT analysis: patients with no detectable bacterial load at baseline were included.
Measure: Number; unit: participants
Arm/Group | CO2 Laser | Traditional Surgery
Number analyzed (Participants) | 10 | 10
participants | 2 | 8

ADVERSE EVENTS:
Time Frame: During procedure and after 1h.
Arm/Group | CO2 Laser | Traditional Surgery
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CO2 Laser (N=10) | Traditional Surgery (N=10)
Bleeding (Injury, poisoning and procedural complications) | 2 (2) | 8 (8)
Pain needing anesthesia (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No